CLINICAL TRIAL: NCT05116631
Title: Analysis of Emergency Department Visits and Activity in Montpellier Dental University Hospital : Study Protocol
Brief Title: Evaluation of Emergency Department Visits and Activity : Study
Acronym: EOTDES
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0649
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-11

CONDITIONS: Dental
Keywords: Dental emergencies; Emergency department; Patients coming to the CHU ADV Montpellier for consultation
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective will be to evaluate the type of care performed and the main reasons for consulting patients for an odontological emergency in order to better adapt to the flow and expectations of patients.

ELIGIBILITY:
Inclusion criteria:

- All adults (>18years) consulting in the emergency department (Montpellier University Hospital)

Exclusion criteria:

* person under 18 years old
* patients who does not speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults (>18years) consulting in the emergency department (Montpellier University Hospital)
Sampling Method: Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of The result for each item of the questionnaire according to the reason for the emergency | 1 day
  The result for each item of the questionnaire according to the reason for the emergency

SECONDARY OUTCOMES:
Number of Participants with Know the type of population received | 1 day
  Know the type of population received, the areas of Montpellier most likely to consult the CSERD, the demand for care

CONTACTS AND LOCATIONS:
Overall Officials: Camille INQUIMBERT, PhD, Study Director — University Hospital, Montpellier; samuel MORAND-MANAS, resident, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC